CLINICAL TRIAL: NCT04168073
Title: Sodium Diet Effect on Aldosterone and Urinary RNA (SALTY)
Acronym: SALTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, J Brian Byrd, MD, MS, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00097366; 1K23HL128909-01A1 (NIH)
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: low sodium diet; high sodium diet; biomarker; aldosterone; mineralocorticoid; mineralocorticoid receptor
MeSH Terms: interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High sodium diet (Experimental)
  Interventions: Other: High-sodium diet 300 mmol sodium/day
- Low sodium diet (Experimental)
  Interventions: Other: Low-sodium diet 10 mmol sodium/day

INTERVENTIONS:
Other: High-sodium diet 300 mmol sodium/day — Day 7 or day 21 high-sodium diet begins for 8 days. Day 15 wash-out begins for 6 days. Pre-made meals for both the high-and low-sodium diet will be provided to each participant by the study team.
  Arms: High sodium diet
Other: Low-sodium diet 10 mmol sodium/day — Day 7 or day 21 low-sodium diet begins for 8 days. Day 15 wash-out begins for 6 days. Pre-made meals for both the high-and low-sodium diet will be provided to each participant by the study team.
  Arms: Low sodium diet

SUMMARY:
This cross-over clinical trial is being conducted to evaluate the difference in urinary messenger RNA (mRNA) biomarkers of mineralocorticoid receptor activation following a low-sodium diet, as compared to a high-sodium diet. The study team will collect urine and blood samples from each participant to study mineralocorticoid receptor-regulated mRNA biomarkers following the consumption of each diet.

The study team will instruct the participants to consume 8 days each of high- (300 mmol/day) and low- (10 mmol/day) sodium meals. The order in which the participants will eat the two study diets will be randomly determined. In between the high- and low-sodium diets, the participants will have a wash-out period of 6 days, during which they will be encouraged to consume their usual diet. Participants will be asked to provide the study team with 24-hour urine samples, random urine samples, and blood samples throughout their participation in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive, as defined by:

  * Systolic blood pressure (SBP) < 140 mmHg and diastolic blood pressure (DBP) < 90 mmHg
  * Never prescribed an antihypertensive medication
* Willingness to refrain from intense exercise (for example, swimming, biking, running)

Exclusion Criteria:

* Hypertension (history of blood pressure ≥ 140/90 mmHg)
* History of hypertensive urgency, hypertensive crisis, or hospitalizations for hypertension
* History of chronic kidney disease
* History of heart failure
* Current food allergy
* Pregnancy
* Known hyperaldosteronism
* Current mineralocorticoid antagonist use
* Current treatment for diabetes mellitus
* Known adrenal insufficiency
* Current glucocorticoid use
* Electrolyte abnormality on baseline laboratory assessment
* Current potassium supplementation
* Urinary tract infection (UTI)
* Significant renal insufficiency or any other condition thought by the Principal Investigator to place the participant at increased risk of injury during the clinical trial or compromise the scientific integrity of the study

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Urinary mineralocorticoid receptor-regulated messenger RNA (mRNA) biomarker | Day 15 (after first diet period)
  Urinary mRNA biomarkers following consumption of a high-sodium and low-sodium diet will be measured using real-time quantitative polymerase chain reaction (RT-qPCR).
Urinary mineralocorticoid receptor-regulated mRNA biomarker | Day 29 (after second diet period)
  Urinary mRNA biomarkers following consumption of a high-sodium and low-sodium diet will be measured using real-time quantitative polymerase chain reaction (RT-qPCR).

SECONDARY OUTCOMES:
Blood pressure | Day 15 (after first diet period)
  Systolic and diastolic blood pressure measurement following consumption of a high-sodium compared to a low-sodium diet
Blood pressure | Day 29 (after second diet period)
  Systolic and diastolic blood pressure measurement following consumption of a high-sodium compared to a low-sodium diet

CONTACTS AND LOCATIONS:
Overall Officials: J Brian Byrd, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
We will de-identify participant information and will share it with a trusted repository, such as National Institutes of Health (NIH) Figshare or The Inter-university Consortium for Political and Social Research (ICPSR).
  We will de-identify and share data obtained from analyzing urinary mRNA biomarkers and measuring the systolic and diastolic blood pressure following consumption of a high-sodium and low-sodium diet. Additionally, specific lab values that support the validity and quality of the study treatment will be shared in a trusted repository.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be deposited into a repository within 1 year of the conclusion of the study.
Access Criteria: No additional access restrictions will be placed on the de-identified data, beyond those required by the repository to access or download the data.

DOCUMENTS (1):
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT04168073/ICF_000.pdf